CLINICAL TRIAL: NCT03032562
Title: Multimodal Measurement of Respiratory Muscle Strength and Function: Validation of Volitional and Non-volitional Tests With Regard to Nocturnal Hypoventilation in Patients With Neuromuscular Disorders and Chronic Obstructive Pulmonary Disease
Brief Title: Respiratory Muscle Strength and Function in Neuromuscular Disorders and Chronic Obstructive Pulmonary Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universität Münster (Other)
Responsible Party: Principal Investigator, Matthias Boentert, MD, Universität Münster
Other Study IDs: KSN_2016_2_MB
Record Dates: First submitted 2017-01-24; First posted 2017-01-26 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2017-01

CONDITIONS: Respiratory Muscle Paralysis
Keywords: respiratory muscle strength; sleep-disordered breathing; neuromuscular disease; chronic-obstructive pulmonary disease
MeSH Terms: conditions — Respiratory Paralysis; Sleep Apnea Syndromes; Neuromuscular Diseases; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1: Patients with neuromuscular disease
  Interventions: Diagnostic Test: Multimodal measurement of respiratory muscle function and strength
- 2: Patients with chronic obstructive pulmonary disease
  Interventions: Diagnostic Test: Multimodal measurement of respiratory muscle function and strength

INTERVENTIONS:
Diagnostic Test: Multimodal measurement of respiratory muscle function and strength — Sleep-studies, capnography, spiromanometry, phrenic nerve conduction studies, magnetic phrenic nerve stimulation, diaphragmatic ultrasound

SUMMARY:
Using an extensive set of both volitional and non-volitional tests of respiratory muscle function and strength it is the aim of this study to

* identify disease-specific patterns of respiratory muscle impairment in different NMD and COPD
* establish which set of tests is predictive of sleep-disordered breathing or daytime hypercapnia in patients with NMD or COPD, respectively.
* to investigate the decline of respiratory muscle function in patients with progressive NMD and COPD along with sleep studies and capnography

DETAILED DESCRIPTION:
Numerous neuromuscular disorders (NMD) are characterized not only by weakness of axial and limb muscles but also by respiratory muscle and upper airway involvement. Respiratory muscle weakness first manifests as sleep-disordered breathing (SDB). SDB in neuromuscular disease mainly comprises alveolar hypoventilation but upper airway collapse may also occur because pharyngeal muscle tone is impaired by both neuromuscular weakness and sleep.

Diaphragmatic weakness and myopathy are hallmarks of advanced obstructive pulmonary disease leading to even greater impairment of gas exchange in affected patients.

Non-invasive ventilation (NIV) should be initiated in patients with diaphragm weakness if significant SDB or hypercapnic respiratory failure is present. Indication criteria for NIV include measurement of spiromanometric parameters such as forced vital capacity (FVC), maximum inspiratory pressure (MIP), or sniff nasal inspiratory pressure (SNIP). These measurements are volitional, i. e. test results are dependent on individual patient effort and may show intraindividual variance which may not properly reflect disease progression or treatment effects, respectively. Associations between volitional and non-volitional methods of respiratory muscle strength testing have been reported mainly for healthy individuals but only scarcely in patients with specific NMD.

Non-volitional tests of respiratory muscle strength include phrenic nerve conduction studies, diaphragmatic ultrasound, and magnetic stimulation of the phrenic nerves in particular. Magnetic stimulation is usually combined with esophageal and gastric manometry yielding the twitch transdiaphragmatic pressure which closely reflects diaphragmatic strength.

It is desirable to obtain validated data on both volitional and non-volitional tests of respiratory muscle strength in various NMD. Validation has to be carried out with regard to both daytime hypercapnia and nocturnal retention of carbon dioxide because the latter often represents the earliest manifestation of respiratory muscle weakness. SDB often starts long before exertional dyspnea or orthopnea develop. Since NIV is one of the mainstays of symptomatic treatment in both NMD and advanced obstructive lung disease, early recognition of SDB is crucial for optimal patient care, and in many conditions, life expectancy and quality of life may be substantially increased by NIV. In this study, FVC, MIP, MEP and SNIP testing along with non-volitional methods and diaphragmatic ultrasound will be applied in order to establish a protocol which may help to reliably predict SDB or need for ventilatory support, respectively.

Patients with chronic obstructive pulmonary disease (COPD) develop flattening, shortening, and weakness of the diaphragm. This is not only due to downward dislocation of the diaphragm but also to impairment of contractile function, tissue structure, and intracellular biochemistry. Respiratory muscle weakness in COPD is of major clinical relevance since maximum inspiratory pressure is an independent predictor of survival in severely affected patients. In addition, hypercapnic respiratory failure due to inspiratory muscle weakness is associated with morbidity and mortality in COPD.

Direct comparison of both volitional and non-volitional measures of respiratory muscle function between patients with diaphragmatic weakness due to neuromuscular disease and patients with COPD is desirable. This approach may allow for further characterization of "impairment patterns" probably specific to either COPD or certain neuromuscular disease, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Patients with NMD (n=100): Amyotrophic lateral sclerosis, Pompe's disease, myotonic dystrophy type 1, limb-girdle muscular dystrophies, spinal muscular atrophy, etc.
* patients with chronic obstructive lung disease (n=100)
* age 18 - 80 years
* written informed consent

Exclusion Criteria:

* significant chest wall deformity
* tracheostomy
* inability to sit in the upright position
* impaired consciousness
* acute or severe medical comorbidity
* mechanical ventilation for more than 4 hours during daytime

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with known neuromuscular disease and individuals with chronic obstructive pulmonary disease (and no neuromuscular disorder)
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2016-12-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-02-28 (Estimated)

PRIMARY OUTCOMES:
Presence of daytime hypercapnia | 1 day
  paCO2 > 45 mmHg
Presence of sleep-disordered breathing | 1 day
  nocturnal tcCO2 > 50 mmHg, delta tcCO2 > 10 mmHg

SECONDARY OUTCOMES:
twitch transdiaphragmatic pressure | 1 day
  difference between intraesophageal and intragastral pressure after posterior magnetic stimulation of the phrenic nerves

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - University Hospital Münster, Department of Sleep Medicine and Neuromuscular Disorders, Münster, North Rhine-Westphalia
  - Bethanien Hospital, Solingen, North Rhine-Westphalia

IPD SHARING:
Plan to Share IPD: No